CLINICAL TRIAL: NCT06422715
Title: Post-transplant Lymphoproliferative Disorders (PTLD): Multicentric Observational Retrospective Cohort Study
Brief Title: PTLD: Multicentric Retrospective Study
Acronym: FIL_PTLD
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Collaborators: Pierre Fabre Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: FIL_PTLD
Record Dates: First submitted 2024-05-07; First posted 2024-05-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: PTLD
Keywords: PTLD; lymphoproliferative disorders; transplant
MeSH Terms: conditions — Lymphoproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with histological diagnosis of PTLD: patients with histological diagnosis obtained from a biopsy sample in 10 years' time frame (from 01/01/2011 to 31/12/2021) of PTLD (from allogeneic transplantation (both SOT and HSCT))

SUMMARY:
This is a multicentric observational retrospective cohort study of patients with histological diagnosis of PTLD.

The aim of the study is to analyze the clinical features and survival of patients who received a PTLD diagnosis with the target to assess a survival outcome, to obtain an epidemiologic and clinical characterization of the subpopulations affected by PTLD, to recognize unfavorable properties, to report the current treatment strategies, to provide rationale for the design of a prospective registry in order to develop future novel treatments.

DETAILED DESCRIPTION:
This is a multicentric observational retrospective cohort study of patients with histological diagnosis of PTLD. Retrospective data will be collected for all cases of PTLD diagnosed during a 10 years period since 1st January 2011 to 31th December 2021.

The following clinical characteristics of the patient at the time of PTLD diagnosis and pathology will be taken into consideration: positivity of EBV virus, serum LDH concentration, PTLD subtype (early lesion, polymorphic or monomorphic PTLD), lymphoma histotype, stage of disease according to the Ann Arbor classification and localization (nodal or extranodal), immunosuppressive regimen taken by the patient since the transplant, therapeutic approach adopted, and response obtained.

ELIGIBILITY:
Inclusion Criteria:

* histological diagnosis of PTLD obtained from a biopsy sample (availability of stocked biopsy sample is requested but not mandatory);
* age over 18 years at time of diagnosis of PTLD;
* previously subjected to allogeneic transplantation (both SOT and HSCT);
* diagnosis of PTLD obtained in 10 years' time frame (from 01/01/2011 to 31/12/2021);
* free and voluntary written informed consent (included unreachable subjects according to Art. 36 UE Regulation 2016/679 and to the current Italian Privacy Regulation).

Exclusion Criteria:

* Patients not meeting the above-mentioned inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will be composed by patients with histological diagnosis of PTLD. The following clinical characteristics of the patient at the diagnosis of PTLD and pathology will be taken into consideration: positivity of EBV virus, serum LDH concentration, PTLD subtype (early lesion, polymorphic or monomorphic PTLD), lymphoma histotype, stage of disease according to the Ann Arbor classification and localization (nodal or extranodal), immunosuppressive regimen taken by the patient since the transplant, therapeutic approach adopted and response obtained.
Sampling Method: Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Overall Survival | from diagnosis of PTLD to patient's death / last FUP - up to 18 months.
  survival after PTLD incidence rating
clinical and epidemiological features | from diagnosis of PTLD to patient's death/ last FUP - up to 18 months.
  analyze the clinical and epidemiological features (e.g. positivity of EBV virus, serum LDH concentration, PTLD subtype (early lesion, polymorphic or monomorphic PTLD), lymphoma histotype, stage of disease according to the Ann Arbor classification and localization (nodal or extranodal), immunosuppressive regimen taken by the patient since the transplant, therapeutic approach adopted and response obtained) of PTLD patients

SECONDARY OUTCOMES:
Rate of Progression Free Survival | from diagnosis of PTLD to patient's death/ last FUP - up to 18 months.
  compare outcomes according to treatment approaches
Overall Response Rate | from treatment of PTLD to patient's death / last FUP - up to 18 months.
  investigate potential treatment effect modifications on outcomes according to patient characteristics
Complete Response Rate to first and subsequent treatments | from treatment of PTLD to patient's death / last FUP - up to 18 months.
  investigate potential treatment effect modifications on outcomes according to patient
Overall Survival stratified by prognostic factors | from diagnosis of PTLD to patient's death/ last FUP - up to 18 months.
  Overall Survival assessment stratified by prognostic factors (EBV, LDH, IPI, age, type of transplant)
Progression Free Survival stratified by prognostic factors | from diagnosis of PTLD to patient's death/ last FUP - up to 18 months.
  Progression Free Survival assessment stratified by prognostic factors (EBV, LDH, IPI, age, type of transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Federica Cavallo, MD, Principal Investigator — Ematologia Universitaria - A.O.U. Citta della Salute e della Scienza di Torino
Locations (21):
- Italy (21):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico - Ematologia, Milan, MI
  - Centro Di Riferimento Oncologico Di Aviano, S.O.C. Oncologia Medica e dei Tumori Immunocorrelati, Aviano
  - Azienda Ospedaliera Papa Giovanni XXIII - Ematologia, Bergamo
  - A.O. UNIVERSITARIA POLICLINICO S.ORSOLA-MALPIGHI DI BOLOGNA - Istituto di Ematologia "Seragnoli", Bologna
  - A.O. Spedali Civili di Brescia - Ematologia, Brescia
  - Ospedale Businco - Divisione di Ematologia, Cagliari
  - A.O. S. Croce e Carle - S.C. di Ematologia e Trapianto di Midollo Osseo, Cuneo
  - A.O. UNIVERSITARIA CAREGGI DI FIRENZE - Unità funzionale di Ematologia, Florence
  - ASST Grande Ospedale Metropolitano Niguarda - SC Ematologia, Miano
  - Istituto Scientifico San Raffaele - Unitа Linfomi - Dipartimento Oncoematologia, Milan
  - AOU Maggiore della Caritа di Novara - SCDU Ematologia, Novara
  - IRCCS ISTITUTO ONCOLOGICO VENETO (IOV) - Oncologia 1, Padua
  - IRCCS Policlinico San Matteo - Divisione di Ematologia, Pavia
  - Policlinico Universitario Campus Bio-Medico - Ematologia - Trapianto cellule staminali - Medicina Trasfusionale e Terapia cellulare, Roma
  - Dipartimento di Medicina Traslazionale e di Precisione - Policlinico Umberto I - Università "La Sapienza" Istituto Ematologia, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Università Cattolica S. Cuore - Ematologia, Roma
  - AOU Senese - U.O.C. Ematologia, Siena
  - A.O. UNIVERSITARIA CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - SC Ematologia, Torino
  - A.O. Città della Salute e della Scienza - Ematologia Universitaria, Torino
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) - SOC Clinica Ematologica, Udine
  - ULSS 8 Berica - Ospedale S. Bortolo - Ematologia, Vicenza